CLINICAL TRIAL: NCT06937255
Title: Validation of Computerized Dynamic Assessment Tasks to Identify the Risk of Developmental Language Disorders (DLD) and Specific Reading Disorder (SRD) in Monolingual and Multilingual Children
Brief Title: Dynamic Assessment of the Risk for Language and Reading Disorders in Monolingual and Multilingual Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 1036
Record Dates: First submitted 2024-03-21; First posted 2025-04-22 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Developmental Dyslexia; Developmental Language Disorder
Keywords: Developmental Dyslexia; Developmental Language Disorder; Dynamic Assessment; computerized assessment; multilingual population; children
MeSH Terms: conditions — Dyslexia; Language Development Disorders

STUDY DESIGN:
Intervention Model Description: The study will compare performance in a parallel manner in two populations: preschool and school-age children.
  Preschool age children will be assessed with the DA screening test for the risk of DLD, whereas school-age children will be assessed with the DA screening test for the risk of SRD. Each of the two groups will be subdivided into 2 groups: typically developing (TD) and atypically developing (AD). Each of the 2 groups will be further subdivided into monolingual and multilingual children. Pairwise comparisons will be performed to assess the capacity of the DA screening tools to discriminate AD from TD children, separately for monolingual and multilingual children.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- TD preschooler, monolingual (Active Comparator): This group will include monolingual children who have not been referred to clinical or educational services for any delay or disorder in language abilities. They will be tested with the MuLiMi battery (lexical, phonological and morphosyntactic tests), including the DA Novel Word Learning Test (NWLT) as DA screening test. Furthermore, they will be assessed with standardized language tests providing benchmark measures for validation.
  Interventions: Diagnostic Test: computerized Dynamic Assessment
- TD preschooler, multilingual (Active Comparator): This group will include multilingual children who have not been referred to clinical or educational services for any delay or disorder in language abilities. They will be tested with the MuLiMi battery (lexical, phonological and morphosyntactic tests), including the DA Novel Word Learning Test (NWLT) as DA screening test. Furthermore, they will be assessed with standardized language tests providing benchmark measures for validation.
  Interventions: Diagnostic Test: computerized Dynamic Assessment
- DLD preschooler, monolingual (Experimental): This group will include monolingual children who have been referred to clinical or educational services because of delays or disorders in language abilities. They will be tested with the MuLiMi battery (lexical, phonological and morphosyntactic tests), including the DA Novel Word Learning Test (NWLT) as DA screening test. Furthermore, they will be assessed with standardized language tests providing benchmark measures for validation.
  Interventions: Diagnostic Test: computerized Dynamic Assessment
- DLD preschooler, multilingual (Experimental): This group will include multilingual children who have been referred to clinical or educational services because of delays or disorders in language abilities. They will be tested with the MuLiMi battery (lexical, phonological and morphosyntactic tests), including the DA Novel Word Learning Test (NWLT) as DA screening test. Furthermore, they will be assessed with standardized language tests providing benchmark measures for validation.
  Interventions: Diagnostic Test: computerized Dynamic Assessment
- TD school-age, monolingual (Active Comparator): This group will include monolingual children who have not been referred to clinical or educational services for any delay or disorder in language abilities. They will be tested with the MuLiMi battery (reading, orthographic and metaphonological tests), including the Dynamic Reading Assessment (DRA) as DA screening test. Furthermore, they will be assessed with standardized reading and language tests providing benchmark measures for validation.
  Interventions: Diagnostic Test: computerized Dynamic Assessment
- TD school-age, multilingual (Active Comparator): This group will include monolingual children who have not been referred to clinical or educational services for any delay or disorder in language abilities. They will be tested with the MuLiMi battery (reading, orthographic and metaphonological tests), including the Dynamic Reading Assessment (DRA) as DA screening test. Furthermore, they will be assessed with standardized reading and language tests providing benchmark measures for validation.
  Interventions: Diagnostic Test: computerized Dynamic Assessment
- SRD school-age, monolingual (Experimental): This group will include monolingual children who have been referred to clinical or educational services for any delay or disorder in language abilities. They will be tested with the MuLiMi battery (reading, orthographic and metaphonological tests), including the Dynamic Reading Assessment (DRA) as DA screening test. Furthermore, they will be assessed with standardized reading and language tests providing benchmark measures for validation.
  Interventions: Diagnostic Test: computerized Dynamic Assessment
- SRD school-age, multilingual (Experimental): This group will include multilingual children who have been referred to clinical or educational services for any delay or disorder in language abilities. They will be tested with the MuLiMi battery (reading, orthographic and metaphonological tests), including the Dynamic Reading Assessment (DRA) as DA screening test. Furthermore, they will be assessed with standardized reading and language tests providing benchmark measures for validation.
  Interventions: Diagnostic Test: computerized Dynamic Assessment

INTERVENTIONS:
Diagnostic Test: computerized Dynamic Assessment — The DA tests (with a duration of about 30 minutes) can be administered by accessing the digital platform MuLiMi, individually with the experimenter or examiner. The tests are in game form and require children to learn the names of characters presented in the context of stories (preschool version) or to learn new codes for reading and writing (primary school version). In both cases, the new materials (names or codes) are repeatedly presented to the child until (s)he reaches an accuracy threshold. The number of repetitions needed to reach the threshold constitutes the main measure of the child's learning capacity, together with the number of errors committed during the various cycles.
  Other Names: MuLiMi Dynamic Assessment tools

SUMMARY:
The project represents the completion of a part of the recently concluded European project MultiMind, in which a computer platform called MuLiMi was developed and validated. The platform hosts screening tests for the identification of the risk of Language and Learning Disorders in preschool and primary school children, respectively. The aim is to validate the Dynamic Assessment (DA) tests (a first test assessing the capacity to learn new words for preschool children and a second one assessing the capacity to learn a new spelling code for school-age children) in a population of monolingual and bilingual children attending preschool and primary school. The main goal of the study is to complete the validation of the two Dynamic Assessment tests implemented in the MuLiMi platform developed for the MultiMind project.

DETAILED DESCRIPTION:
Dynamic Assessment tests are characterized by their emphasis on the learning process activated during the test itself, focusing on measuring the improvement achieved from the beginning to the end of the test rather than the absolute level of performance. They are thus considered measures of the learning potential (in this case, language and spelling) of the assessed subject. This type of testing is used as an integration of static assessment (traditional, aimed at detecting absolute performance level) and has proven particularly useful in the assessment of multilingual children.

However, computerized tests that can also be used remotely are not currently available. For these reasons, it was found particularly useful to include this type of task within the MuLiMi computerized battery. While the other tests hosted on the MuLiMi platform concern specific L1-L2 pairs, DA tests can be applied regardless of the L1 (provided a minimum L2 mastery is present so as to understand the requests) because they assess the capacity to learn new information and are thus rather independent of previous knowledge. This study will provide baseline data for the MuLiMi battery applied to children belonging to any language minority group and thus enable it to be used comprehensively in the future for the purpose of risk assessment of language and learning disorders.

ELIGIBILITY:
Inclusion Criteria:

* age 4-6 years (Kindergarten) or 7-9 years (Primary school);
* Attendance at an Italian-language school in Italy or Switzerland/Germany.

Additional inclusion criteria for the multilingual group only:

* (i) At least one parent speaks at least one language other than Italian in the family;
* (ii) Continuous exposure to the Italian language for at least two years.

Exclusion Criteria:

* Intellectual disability, major psychopathological disorders, exposure to Italian language for less than two years.

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2023-04-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
accuracy during task performance | one or two days (one or two consecutive sessions depending on participant's age, collaboration and fatigue)
  total number and % correct answers, number and % errors during task performance
efficiency during task performance | Intervention occurs during assessment: assessment will last one or two days (one or two consecutive sessions depending on participant's age, collaboration and fatigue)
  number of repeated cycles, number of cycles needed to reach target performance

CONTACTS AND LOCATIONS:
Overall Officials: Maria Luisa Lorusso, Ph.D, Principal Investigator — IRCCS E. Medea
Locations (1):
- IRCCS E. Medea, polo di Bosisio Parini, Bosisio Parini, LC, Italy

REFERENCES:
- [Background] MacLeod AAN, Glaspey AM. Dynamic assessment of multilingual children's word learning. Int J Lang Commun Disord. 2022 Jul;57(4):822-851. doi: 10.1111/1460-6984.12723. Epub 2022 Apr 16. PMID 35429340
- [Background] Orellana CI, Wada R, Gillam RB. The Use of Dynamic Assessment for the Diagnosis of Language Disorders in Bilingual Children: A Meta-Analysis. Am J Speech Lang Pathol. 2019 Aug 9;28(3):1298-1317. doi: 10.1044/2019_AJSLP-18-0202. Epub 2019 Jun 13. PMID 31194570
- [Background] Hunt E, Nang C, Meldrum S, Armstrong E. Can Dynamic Assessment Identify Language Disorder in Multilingual Children? Clinical Applications From a Systematic Review. Lang Speech Hear Serv Sch. 2022 Apr 11;53(2):598-625. doi: 10.1044/2021_LSHSS-21-00094. Epub 2022 Mar 1. PMID 35230888